CLINICAL TRIAL: NCT05199311
Title: A Phase I/II Study of Carfilzomib, Iberdomide (CC-220) and Dexamethasone (KID) in Patients With Newly Diagnosed Transplant Eligible Multiple Myeloma
Brief Title: Carfilzomib, Iberdomide (CC-220) and Dexamethasone (KID) in Transplant Eligible Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2021-0842
Record Dates: First submitted 2021-11-03; First posted 2022-01-20 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; iberdomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Starting Dose -1 (Experimental): CC-220/Iberdomide: 1.1 mg [CC-220 dosing schedule: daily for 21 days of each 28-day cycle]
  Carfilzomib: 20 mg/m2 C1D1 56 mg/m2 thereafter [Days 1, 8, 15 per 28-day cycle]
  Dexamethasone: 40 mg (≤ 75 years) 20 mg (> 75 years) [Days 1, 8, 15, 22 per 28-day cycle]
  Treatment will continue with carfilzomib, iberdomide, and dexamethasone for up to 4 cycles (28 days) at the physician's discretion followed by the Autologous Stem Cell Transplant. Patients will be followed every 3 months for up to 2 years, or until PD or the start of a new line of therapy.
  Interventions: Drug: Carfilzomib; Drug: Iberdomide; Drug: Oral Dexamethasone
- Dose Level 1 (Experimental): CC-220/Iberdomide: 1.3 mg [CC-220 dosing schedule: daily for 21 days of each 28-day cycle]
  Carfilzomib: 20 mg/m2 C1D1 56 mg/m2 thereafter [Days 1, 8, 15 per 28-day cycle]
  CC-220 dose level 1 enrollment will occur following an independent safety review two months after the first 10 patients have completed at least 2 cycles of therapy at dose level -1.
  Dexamethasone: 40 mg (≤ 75 years) 20 mg (> 75 years) [Days 1, 8, 15, 22 per 28-day cycle]
  Treatment will continue with carfilzomib, iberdomide, and dexamethasone for up to 4 cycles (28 days) at the physician's discretion followed by the Autologous Stem Cell Transplant. Patients will be followed every 3 months for up to 2 years, or until PD or the start of a new line of therapy.
  Interventions: Drug: Carfilzomib; Drug: Iberdomide; Drug: Oral Dexamethasone
- Dose Level 2 (Experimental): CC-220/Iberdomide: 1.6 mg [CC-220 dosing schedule: daily for 21 days of each 28-day cycle]
  Carfilzomib: 20 mg/m2 C1D1 56 mg/m2 thereafter [Days 1, 8, 15 per 28-day cycle]
  CC-220 dose level 2 enrollment will occur following an independent safety review two months after the first 10 patients have completed at least 2 cycles of therapy at dose level 1.
  Dexamethasone: 40 mg (≤ 75 years) 20 mg (> 75 years) [Days 1, 8, 15, 22 per 28-day cycle]
  Treatment will continue with carfilzomib, iberdomide, and dexamethasone for up to 4 cycles (28 days) at the physician's discretion followed by the Autologous Stem Cell Transplant. Patients will be followed every 3 months for up to 2 years, or until PD or the start of a new line of therapy.
  Interventions: Drug: Carfilzomib; Drug: Iberdomide; Drug: Oral Dexamethasone
- Dose Level -2 (Experimental): CC-220/Iberdomide: 0.75 mg [CC-220 dosing schedule: daily for 21 days of each 28-day cycle]
  Carfilzomib: 20 mg/m2 C1D1 56 mg/m2 thereafter [Days 1, 8, 15 per 28-day cycle]
  Dexamethasone: 40 mg (≤ 75 years) 20 mg (> 75 years) [Days 1, 8, 15, 22 per 28-day cycle]
  Treatment will continue with carfilzomib, iberdomide, and dexamethasone for up to 4 cycles (28 days) at the physician's discretion followed by the Autologous Stem Cell Transplant. Patients will be followed every 3 months for up to 2 years, or until PD or the start of a new line of therapy.
  Interventions: Drug: Carfilzomib; Drug: Iberdomide; Drug: Oral Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — 20 mg/m2 C1D1; 56 mg/m2 thereafter
Drug: Iberdomide — Oral CC-220 at dose specified by cohort dose level from Day 1-21 of each 28-day cycle
Drug: Oral Dexamethasone — 40 mg (<=75 years old); 20 mg (>75 years old)

SUMMARY:
This is a multi-institution, open label, phase I/II study of Iberdomide, Carfilzomib, and dexamethasone (KID) in patients with newly diagnosed transplant eligible MM.

DETAILED DESCRIPTION:
This is a multi-institution, open label, phase I/II study of Iberdomide, Carfilzomib, and dexamethasone (KID) in patients with newly diagnosed transplant eligible MM.

As part of a dose escalation phase, the first 10 patients will be enrolled at dose level -1 (Iberdomide 1.1 mg po daily days 1-21). Two months after the first 10 patients have completed at least 2 cycles of therapy in dose level -1, an Independent Safety Review Committee will review the safety data. Assuming the combination is determined to have adequate safety and tolerability, 10 patients will be enrolled at dose level 1 (Iberdomide 1.3 mg po daily days 1-21). After an independent safety review two months after 10 patients have completed at least 2 cycles of therapy in dose level 1, the remaining 46 patients will be enrolled at dose level 2 (Iberdomide 1.6 mg po daily days 1-21).

Treatment will continue for up to 4 cycles (28 days) at the physician's discretion followed by the Autologous Stem Cell Transplant. Patients will be followed every 3 months for up to 2 years, or until disease progression or the start of a new line of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Documented newly diagnosed multiple myeloma

   a. At least 25% of patients accrued should be high risk as defined by IMWG or mSMART criteria.
2. Patient should be deemed transplant eligible.
3. Patients may not have had more than 1 cycle of prior induction therapy. If a patient has had 1 cycle of prior multiple myeloma therapy, the patient must have had documented measurable disease prior to initiation of cycle 1.
4. Subjects must satisfy the following criteria to be enrolled in the study:

   1. Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF).
   2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
   3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
5. Subjects must have a documented diagnosis of MM and have measurable disease defined as:

   1. M-protein (serum and/or urine protein electrophoresis (sPEP or uPEP)): sPEP≥0.5 g/dL or uPEP ≥ 200 mg/24 hours and/or
   2. Light chain MM without measurable disease in the serum or urine: serum immunoglobulin free light chain ≥ 10 mg/dL (100 mg/L) and abnormal serum immunoglobulin kappa lambda free light chain ratio
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2.
7. A female of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral salpingectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months) and must:

   a. Have two negative pregnancy tests as verified by the Investigator prior to starting study treatment. She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence from heterosexual contact.
8. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with two forms of contraception: one highly effective, and one additional effective (barrier) measure of contraception without interruption 28 days prior to starting investigational product, during the study treatment (including dose interruptions), and for at least 28 days after the last dose of iberdomide.
9. Male subjects must:

   a. Male subjects must practice complete abstinence (True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence [e.g. calendar, ovulation, symptothermal or post-ovulation methods] and withdrawal are not acceptable methods of contraception.) or agree to use a condom during sexual contact with a pregnant female or a FCBP while taking iberdomide, during dose interruptions and for at least 28 days following the last dose of iberdomide even he has undergone a successful vasectomy.
10. Males must agree to refrain from donating sperm while on study treatment, during dose interruptions and for at least 28 days following last dose of study treatment.
11. All subjects must agree to refrain from donating blood while on study treatment, during dose interruptions and for at least 28 days following the last dose of study treatment.
12. All male and female subjects must follow all requirements defined in the Pregnancy Prevention Program.

Note: A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

Exclusion Criteria:

1. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
3. Subject has any condition that confounds the ability to interpret data from the study
4. Subject has nonsecretory multiple myeloma
5. Subjects with Plasma Cell leukemia or amyloidosis (with the exception of isolated marrow involvement).
6. Any of the following laboratory abnormalities:

   1. Absolute neutrophil count (ANC) < 1,000/μL
   2. Platelet count < 50,000/μL. It is not permissible to transfuse subjects to achieve minimum platelet counts.
   3. Corrected serum calcium > 13.5 mg/dL (> 3.4 mmol/L)
   4. Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) or serum glutamic pyruvic transaminase (SGPT)/alanine aminotransferase (ALT) ≥ 2.5 x upper limit of normal (ULN)
   5. Serum total bilirubin, direct bilirubin, or alkaline phosphatase ≥ 1.5 x ULN
   6. Subjects with serious renal impairment ([CrCl] < 30 mL/min) or requiring dialysis would be excluded
7. Subjects with peripheral neuropathy ≥ Grade 2
8. Subjects with gastrointestinal disease that may significantly alter the absorption of iberdomide
9. Subjects with a prior history of malignancies, other than MM, unless the subject has been free of the disease for ≥ 3 years with the exception of the following noninvasive malignancies:

   1. Basal cell carcinoma of the skin
   2. Squamous cell carcinoma of the skin
   3. Carcinoma in situ of the cervix
   4. Carcinoma in situ of the breast
   5. Incidental histological findings of prostate cancer such as T1a or T1b using the Tumor/Node/Metastasis (TNM) classification of malignant tumors or prostate cancer that is curative
10. Subject has a history of anaphylaxis or hypersensitivity to thalidomide, lenalidomide, or pomalidomide
11. Contraindications to the other treatment regimens, as per local prescribing information
12. Subject has received any of the following within the last 14 days of initiating IP:

    1. Plasmapheresis
    2. Major surgery (as defined by the Investigator)
    3. Radiation therapy other than local therapy for MM associated bone lesions
    4. Use of any systemic myeloma drug therapy
13. Subject has been treated with an investigational agent (ie, an agent not commercially available) within 28 days or 5 half-lives (whichever is longer) of initiating IP
14. Subject has any one of the following:

    1. Active congestive heart failure (New York Heart Association Class III to IV), symptomatic ischemia, uncontrolled arrhythmias, screening ECG with corrected QT interval (QTc) of > 470 msec, pericardial disease, or myocardial infarction within 4 months prior to randomization.
    2. Unstable or poorly controlled angina pectoris, including the Prinzmetal variant of angina pectoris
    3. Subject experienced a cardiac event within 6 months prior to the first dose of IP
15. Subject has current or prior use of immunosuppressive medication within 14 days prior to the first dose of IP. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical or local steroid injections (eg, intra-articular injection)
    2. Glucocorticoid therapy within 14 days prior to randomization that exceeds a cumulative dose of 160 mg of dexamethasone or equivalent dose of other corticosteroids.
    3. Steroids as premedication for hypersensitivity reactions (eg, computed tomography [CT] scan premedication)
16. Subject has taken a strong inhibitor or inducer of CYP3A4/5 including grapefruit, St. John's Wort or related products within two weeks prior to dosing and during the course of study
17. Subject known to test positive for human immunodeficiency virus (HIV), uncontrolled or active viral hepatitis.
18. Subject is unable or unwilling to undergo protocol required thromboembolism prophylaxis
19. Subject is a female who is pregnant, nursing or breastfeeding, or who intends to become pregnant during the participation in the study, or who will not agree to comply with contraceptive requirements or pregnancy monitoring requirements
20. Left ventricular ejection fraction (LVEF) < 40% as determined by echocardiogram (ECHO)
21. Prior use of iberdomide
22. Subject is pregnant
23. Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment. Uncontrolled hypertension is defined as: a subject whose blood pressure exceeds ≥ 160 mmHg systolic or ≥ 100 mmHg diastolic when taken in accordance with the European Society of Hypertension/European Society of Cardiology 2018 guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of treatment emergent adverse events (TEAEs) | Measured after cycle 4 of induction KID (each cycle is 28 days)
  Rate of patients with treatment emergent adverse events (TEAEs) overall and per dose level
CR and sCR | Measured after cycle 4 of induction KID (each cycle is 28 days)
  Evaluation of the rate of complete remission (CR) + stringent complete (sCR) remission for patients receiving 2-4 cycles of the combination of KID followed by ASCT in patients with newly diagnosed MM.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Participants will be followed for response assessment every 28 days until progression of disease or a subsequent myeloma regimen has been started. On treatment study duration will last up to 12 months; Post treatment follow up will last up to two years.
  Assessment of overall response rate (ORR) of newly diagnosed transplant-eligible MM patients.
Progression Free Survival (PFS) | Participants will be followed for response assessment every 28 days until progression of disease or a subsequent myeloma regimen has been started. On treatment study duration will last up to 12 months; Post treatment follow up will last up to two years.
  Assessment of progression-free survival (PFS) of newly diagnosed transplant-eligible MM patients.
Overall Survival (OS) | Participants will be followed for response assessment every 28 days until progression of disease or a subsequent myeloma regimen has been started. On treatment study duration will last up to 12 months; Post treatment follow up will last up to two years.
  Assessment of overall survival (OS) of newly diagnosed transplant-eligible MM patients.

CONTACTS AND LOCATIONS:
Overall Officials: Noa Biran, MD, Principal Investigator — Hackensack Meridian Health
Locations (2):
- United States (2):
  - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - John Theurer Cancer Center, Hackensack, New Jersey

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Agarwal A, Chow E, Bhutani M, Voorhees PM, Friend R, Usmani SZ. Practical Considerations in Managing Relapsed Multiple Myeloma. Clin Lymphoma Myeloma Leuk. 2017 Feb;17(2):69-77. doi: 10.1016/j.clml.2016.11.010. Epub 2016 Nov 23. PMID 27986429
- [Background] Ali SA, Shi V, Maric I, Wang M, Stroncek DF, Rose JJ, Brudno JN, Stetler-Stevenson M, Feldman SA, Hansen BG, Fellowes VS, Hakim FT, Gress RE, Kochenderfer JN. T cells expressing an anti-B-cell maturation antigen chimeric antigen receptor cause remissions of multiple myeloma. Blood. 2016 Sep 29;128(13):1688-700. doi: 10.1182/blood-2016-04-711903. Epub 2016 Jul 13. PMID 27412889
- [Background] Amatangelo M, Bjorklund CC, Kang J, Polonskaia A, Viswanatha S, Thakurta A. Iberdomide (CC-220) has Synergistic Anti-Multiple Myeloma Activity in Combination with both Bortezomib and Dexamethasone, or in combination with Daratumumab in vitro. Blood. 2018;132(Suppl 1):1935.
- [Background] Avet-Loiseau H, Casneuf T, Chiu C, Laubach J, Lee J, Moreau P, et al. Evaluation of Minimal Residual Disease (MRD) in Relapsed/Refractory Multiple Myeloma (RRMM) Patients Treated with Daratumumab in Combination with Lenalidomide Plus Dexamethasone or Bortezomib Plus Dexamethasone. Blood. 2016; 128(22):246.
- [Background] Benboubker L, Dimopoulos MA, Dispenzieri A, Catalano J, Belch AR, Cavo M, Pinto A, Weisel K, Ludwig H, Bahlis N, Banos A, Tiab M, Delforge M, Cavenagh J, Geraldes C, Lee JJ, Chen C, Oriol A, de la Rubia J, Qiu L, White DJ, Binder D, Anderson K, Fermand JP, Moreau P, Attal M, Knight R, Chen G, Van Oostendorp J, Jacques C, Ervin-Haynes A, Avet-Loiseau H, Hulin C, Facon T; FIRST Trial Team. Lenalidomide and dexamethasone in transplant-ineligible patients with myeloma. N Engl J Med. 2014 Sep 4;371(10):906-17. doi: 10.1056/NEJMoa1402551. PMID 25184863
- [Background] Berdeja J, Lin Y, Raje N, Munshi N, Siegel D, Liedtke M, et al. Durable Clinical Responses in Heavily Pretreated Patients with Relapsed/Refractory Multiple Myeloma: Updated Results from a Multicenter Study of bb2121 Anti-Bcma CAR T Cell Therapy. Blood. 2017; 130 (Suppl 1): 740.
- [Background] Biran N, Siegel D, Berdeja JG, Raje N, Cornell RF, Alsina M, Kovacsovics T, Fang B, Kimball AS, Landgren O. Weekly carfilzomib, lenalidomide, and dexamethasone in relapsed or refractory multiple myeloma: A phase 1b study. Am J Hematol. 2019 Jul;94(7):794-802. doi: 10.1002/ajh.25498. Epub 2019 May 13. PMID 31021005
- [Background] Bjorklund C, Kang J, Lu L, Amatangelo M, Chiu H, Hagner P, et al. CC-122 Is a Cereblon Modulating Agent That Is Active in Lenalidomide-Resistant and Lenalidomide/DexamethasoneDouble-Resistant Multiple Myeloma Pre-Clinical Models. Blood. 2016;128(Suppl 1):1592.
- [Background] Botta C, Ciliberto D, Rossi M, Staropoli N, Cuce M, Galeano T, Tagliaferri P, Tassone P. Network meta-analysis of randomized trials in multiple myeloma: efficacy and safety in relapsed/refractory patients. Blood Adv. 2017 Feb 27;1(7):455-466. doi: 10.1182/bloodadvances.2016003905. eCollection 2017 Feb 28. PMID 29296961
- [Background] Brudno JN, Maric I, Hartman SD, Rose JJ, Wang M, Lam N, Stetler-Stevenson M, Salem D, Yuan C, Pavletic S, Kanakry JA, Ali SA, Mikkilineni L, Feldman SA, Stroncek DF, Hansen BG, Lawrence J, Patel R, Hakim F, Gress RE, Kochenderfer JN. T Cells Genetically Modified to Express an Anti-B-Cell Maturation Antigen Chimeric Antigen Receptor Cause Remissions of Poor-Prognosis Relapsed Multiple Myeloma. J Clin Oncol. 2018 Aug 1;36(22):2267-2280. doi: 10.1200/JCO.2018.77.8084. Epub 2018 May 29. PMID 29812997
- [Background] Chari A, Rodriguez-Otero P, McCarthy H, Suzuki K, Hungria V, Sureda Balari A, Perrot A, Hulin C, Magen H, Iida S, Maisnar V, Karlin L, Pour L, Parasrampuria DA, Masterson T, Kosh M, Yang S, Delioukina M, Qi M, Carson R, Touzeau C. Subcutaneous daratumumab plus standard treatment regimens in patients with multiple myeloma across lines of therapy (PLEIADES): an open-label Phase II study. Br J Haematol. 2021 Mar;192(5):869-878. doi: 10.1111/bjh.16980. Epub 2020 Jul 30. PMID 33216361
- [Background] Cowan AJ, Allen C, Barac A, Basaleem H, Bensenor I, Curado MP, Foreman K, Gupta R, Harvey J, Hosgood HD, Jakovljevic M, Khader Y, Linn S, Lad D, Mantovani L, Nong VM, Mokdad A, Naghavi M, Postma M, Roshandel G, Shackelford K, Sisay M, Nguyen CT, Tran TT, Xuan BT, Ukwaja KN, Vollset SE, Weiderpass E, Libby EN, Fitzmaurice C. Global Burden of Multiple Myeloma: A Systematic Analysis for the Global Burden of Disease Study 2016. JAMA Oncol. 2018 Sep 1;4(9):1221-1227. doi: 10.1001/jamaoncol.2018.2128. PMID 29800065
- [Background] Cho SF, Anderson KC, Tai YT. Targeting B Cell Maturation Antigen (BCMA) in Multiple Myeloma: Potential Uses of BCMA-Based Immunotherapy. Front Immunol. 2018 Aug 10;9:1821. doi: 10.3389/fimmu.2018.01821. eCollection 2018. PMID 30147690
- [Background] Darzalex. [Package Insert]. Horsham, PA: Janssen Biotech. Available from: https://www.janssenmd.com/pdf/darzalex/darzalex_pi.pdf.
- [Background] Darzalex. [Summary of Product Characteristics]. Available from: https://www.ema.europa.eu/en/documents/product-information/darzalex-epar-product- information_en.pdf
- [Background] Darzalex FASPRO. [Package Insert]. Horsham, PA: Janssen Biotech. Available from: http://www.janssenlabels.com/package-insert/product-monograph/prescribing- information/DARZALEX+Faspro-pi.pdf.
- [Background] Darzalex FASPRO. [Summary of Product Characteristics]. Available from: https://www.ema.europa.eu/en/documents/product-information/darzalex-epar-product- information_en.pdf
- [Background] Davies FE, Raje N, Hideshima T, Lentzsch S, Young G, Tai YT, Lin B, Podar K, Gupta D, Chauhan D, Treon SP, Richardson PG, Schlossman RL, Morgan GJ, Muller GW, Stirling DI, Anderson KC. Thalidomide and immunomodulatory derivatives augment natural killer cell cytotoxicity in multiple myeloma. Blood. 2001 Jul 1;98(1):210-6. doi: 10.1182/blood.v98.1.210. PMID 11418482
- [Background] Deaglio S, Vaisitti T, Billington R, Bergui L, Omede' P, Genazzani AA, Malavasi F. CD38/CD19: a lipid raft-dependent signaling complex in human B cells. Blood. 2007 Jun 15;109(12):5390-8. doi: 10.1182/blood-2006-12-061812. Epub 2007 Feb 27. PMID 17327405
- [Background] Dimopoulos MA, Moreau P, Palumbo A, Joshua D, Pour L, Hajek R, Facon T, Ludwig H, Oriol A, Goldschmidt H, Rosinol L, Straub J, Suvorov A, Araujo C, Rimashevskaya E, Pika T, Gaidano G, Weisel K, Goranova-Marinova V, Schwarer A, Minuk L, Masszi T, Karamanesht I, Offidani M, Hungria V, Spencer A, Orlowski RZ, Gillenwater HH, Mohamed N, Feng S, Chng WJ; ENDEAVOR Investigators. Carfilzomib and dexamethasone versus bortezomib and dexamethasone for patients with relapsed or refractory multiple myeloma (ENDEAVOR): a randomised, phase 3, open-label, multicentre study. Lancet Oncol. 2016 Jan;17(1):27-38. doi: 10.1016/S1470-2045(15)00464-7. Epub 2015 Dec 5. PMID 26671818
- [Background] Dimopoulos M, White D, Benboubker L, Cook G, Leiba M, Morton J, et al. Daratumumab, Lenalidomide, and Dexamethasone (DRd) Versus Lenalidomide and Dexamethasone (Rd) in Relapsed or Refractory Multiple Myeloma (RRMM): Updated Efficacy and Safety Analysis of Pollux. Blood. 2017;130(Suppl 1):739.
- [Background] Dimopoulos MA, Oriol A, Nahi H, San-Miguel J, Bahlis NJ, Usmani SZ, Rabin N, Orlowski RZ, Komarnicki M, Suzuki K, Plesner T, Yoon SS, Ben Yehuda D, Richardson PG, Goldschmidt H, Reece D, Lisby S, Khokhar NZ, O'Rourke L, Chiu C, Qin X, Guckert M, Ahmadi T, Moreau P; POLLUX Investigators. Daratumumab, Lenalidomide, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2016 Oct 6;375(14):1319-1331. doi: 10.1056/NEJMoa1607751. PMID 27705267
- [Background] Durie BGM, Hoering A, Abidi MH, Rajkumar SV, Epstein J, Kahanic SP, Thakuri M, Reu F, Reynolds CM, Sexton R, Orlowski RZ, Barlogie B, Dispenzieri A. Bortezomib with lenalidomide and dexamethasone versus lenalidomide and dexamethasone alone in patients with newly diagnosed myeloma without intent for immediate autologous stem-cell transplant (SWOG S0777): a randomised, open-label, phase 3 trial. Lancet. 2017 Feb 4;389(10068):519-527. doi: 10.1016/S0140-6736(16)31594-X. Epub 2016 Dec 23. PMID 28017406
- [Background] Durie BGM, Hoering A, Sexton R, Abidi MH, Epstein J, Rajkumar SV, Dispenzieri A, Kahanic SP, Thakuri MC, Reu FJ, Reynolds CM, Orlowski RZ, Barlogie B. Longer term follow-up of the randomized phase III trial SWOG S0777: bortezomib, lenalidomide and dexamethasone vs. lenalidomide and dexamethasone in patients (Pts) with previously untreated multiple myeloma without an intent for immediate autologous stem cell transplant (ASCT). Blood Cancer J. 2020 May 11;10(5):53. doi: 10.1038/s41408-020-0311-8. PMID 32393732
- [Background] Engelhardt M, Terpos E, Kleber M, Gay F, Wasch R, Morgan G, Cavo M, van de Donk N, Beilhack A, Bruno B, Johnsen HE, Hajek R, Driessen C, Ludwig H, Beksac M, Boccadoro M, Straka C, Brighen S, Gramatzki M, Larocca A, Lokhorst H, Magarotto V, Morabito F, Dimopoulos MA, Einsele H, Sonneveld P, Palumbo A; European Myeloma Network. European Myeloma Network recommendations on the evaluation and treatment of newly diagnosed patients with multiple myeloma. Haematologica. 2014 Feb;99(2):232-42. doi: 10.3324/haematol.2013.099358. PMID 24497560
- [Background] Facon T, Lonial S, Weiss B, Suvannasankha A, Fay JW, Arnulf B, et al. Daratumumab in Combination with Pomalidomide and Dexamethasone for Relapsed and/or Refractory Multiple Myeloma (RRMM) Patients with >/=2 Prior Lines of Therapy: Updated Analysis of MMY1001. Blood. 2017;130(Suppl 1):1824.
- [Background] Facon T, Dimopoulos MA, Dispenzieri A, Catalano JV, Belch A, Cavo M, Pinto A, Weisel K, Ludwig H, Bahlis NJ, Banos A, Tiab M, Delforge M, Cavenagh JD, Geraldes C, Lee JJ, Chen C, Oriol A, De La Rubia J, White D, Binder D, Lu J, Anderson KC, Moreau P, Attal M, Perrot A, Arnulf B, Qiu L, Roussel M, Boyle E, Manier S, Mohty M, Avet-Loiseau H, Leleu X, Ervin-Haynes A, Chen G, Houck V, Benboubker L, Hulin C. Final analysis of survival outcomes in the phase 3 FIRST trial of up-front treatment for multiple myeloma. Blood. 2018 Jan 18;131(3):301-310. doi: 10.1182/blood-2017-07-795047. Epub 2017 Nov 17. PMID 29150421
- [Background] Fonseca R, Bergsagel PL, Drach J, Shaughnessy J, Gutierrez N, Stewart AK, Morgan G, Van Ness B, Chesi M, Minvielle S, Neri A, Barlogie B, Kuehl WM, Liebisch P, Davies F, Chen-Kiang S, Durie BG, Carrasco R, Sezer O, Reiman T, Pilarski L, Avet-Loiseau H; International Myeloma Working Group. International Myeloma Working Group molecular classification of multiple myeloma: spotlight review. Leukemia. 2009 Dec;23(12):2210-21. doi: 10.1038/leu.2009.174. Epub 2009 Oct 1. PMID 19798094
- [Background] Fraietta JA, Lacey SF, Orlando EJ, Pruteanu-Malinici I, Gohil M, Lundh S, Boesteanu AC, Wang Y, O'Connor RS, Hwang WT, Pequignot E, Ambrose DE, Zhang C, Wilcox N, Bedoya F, Dorfmeier C, Chen F, Tian L, Parakandi H, Gupta M, Young RM, Johnson FB, Kulikovskaya I, Liu L, Xu J, Kassim SH, Davis MM, Levine BL, Frey NV, Siegel DL, Huang AC, Wherry EJ, Bitter H, Brogdon JL, Porter DL, June CH, Melenhorst JJ. Determinants of response and resistance to CD19 chimeric antigen receptor (CAR) T cell therapy of chronic lymphocytic leukemia. Nat Med. 2018 May;24(5):563-571. doi: 10.1038/s41591-018-0010-1. Epub 2018 Apr 30. PMID 29713085
- [Background] Gay F, et al. Efficacy of carfilzomib lenalidomide dexamethasone (KRd) with or without transplantation in newly diagnosed myeloma according to risk status: results from the FORTE trial. J. Clin. Oncol. 2019;37(no. 15_suppl):8002
- [Background] Gorgun G, Calabrese E, Soydan E, Hideshima T, Perrone G, Bandi M, Cirstea D, Santo L, Hu Y, Tai YT, Nahar S, Mimura N, Fabre C, Raje N, Munshi N, Richardson P, Anderson KC. Immunomodulatory effects of lenalidomide and pomalidomide on interaction of tumor and bone marrow accessory cells in multiple myeloma. Blood. 2010 Oct 28;116(17):3227-37. doi: 10.1182/blood-2010-04-279893. Epub 2010 Jul 22. PMID 20651070
- [Background] Gandhi AK, Kang J, Capone L, Parton A, Wu L, Zhang LH, Mendy D, Lopez-Girona A, Tran T, Sapinoso L, Fang W, Xu S, Hampton G, Bartlett JB, Schafer P. Dexamethasone synergizes with lenalidomide to inhibit multiple myeloma tumor growth, but reduces lenalidomide-induced immunomodulation of T and NK cell function. Curr Cancer Drug Targets. 2010 Mar;10(2):155-67. doi: 10.2174/156800910791054239. PMID 20088798
- [Background] Gandhi AK, Kang J, Havens CG, Conklin T, Ning Y, Wu L, Ito T, Ando H, Waldman MF, Thakurta A, Klippel A, Handa H, Daniel TO, Schafer PH, Chopra R. Immunomodulatory agents lenalidomide and pomalidomide co-stimulate T cells by inducing degradation of T cell repressors Ikaros and Aiolos via modulation of the E3 ubiquitin ligase complex CRL4(CRBN.). Br J Haematol. 2014 Mar;164(6):811-21. doi: 10.1111/bjh.12708. Epub 2013 Dec 13. PMID 24328678
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Howlader N, Noone AM, Krapcho M, Miller D, Bishop K, Altekruse SF, et al. SEER Cancer Statistics Review (CSR), 1975-2013, National Cancer Institute. Bethesda, MD, https://seer.cancer.gov/archive/csr/1975_2013/, based on November 2015 SEER data submission, posted to the SEER web site, April 2016.
- [Background] Hoy SM. Carfilzomib Triple Combination Therapy: A Review in Relapsed Multiple Myeloma. Target Oncol. 2016 Apr;11(2):255-62. doi: 10.1007/s11523-016-0428-7. PMID 26972294
- [Background] Imnovid. [Summary of Product Characteristics]. Uxbridge, United Kingdom: Celgene Europe Ltd. Available from: http://www.ema.europa.eu/docs/en_GB/document_library/EPAR_- _Product_Information/human/002682/WC500147717.pdf.
- [Background] Ito T, Ando H, Suzuki T, Ogura T, Hotta K, Imamura Y, Yamaguchi Y, Handa H. Identification of a primary target of thalidomide teratogenicity. Science. 2010 Mar 12;327(5971):1345-50. doi: 10.1126/science.1177319. PMID 20223979
- [Background] Jennison C, Turnbull BW. Group Sequential Methods with Applications to Clinical Trials. 1st ed. Boca Raton, FL: CRC Chapman & Hall; c1999.
- [Background] John LB, Ward AC. The Ikaros gene family: transcriptional regulators of hematopoiesis and immunity. Mol Immunol. 2011 May;48(9-10):1272-8. doi: 10.1016/j.molimm.2011.03.006. Epub 2011 Apr 7. PMID 21477865
- [Background] Katz M, Bjorklund CC, Thakurta A, Serbina N. Mechanistic insights of pomalidomide activity in combination with bortezomib and dexamethasone in multiple myeloma and immune cells. Blood. 2018;132(suppl 1):1934.
- [Background] Kronke J, Udeshi ND, Narla A, Grauman P, Hurst SN, McConkey M, Svinkina T, Heckl D, Comer E, Li X, Ciarlo C, Hartman E, Munshi N, Schenone M, Schreiber SL, Carr SA, Ebert BL. Lenalidomide causes selective degradation of IKZF1 and IKZF3 in multiple myeloma cells. Science. 2014 Jan 17;343(6168):301-5. doi: 10.1126/science.1244851. Epub 2013 Nov 29. PMID 24292625
- [Background] Kumar SK, Lee JH, Lahuerta JJ, Morgan G, Richardson PG, Crowley J, Haessler J, Feather J, Hoering A, Moreau P, LeLeu X, Hulin C, Klein SK, Sonneveld P, Siegel D, Blade J, Goldschmidt H, Jagannath S, Miguel JS, Orlowski R, Palumbo A, Sezer O, Rajkumar SV, Durie BG; International Myeloma Working Group. Risk of progression and survival in multiple myeloma relapsing after therapy with IMiDs and bortezomib: a multicenter international myeloma working group study. Leukemia. 2012 Jan;26(1):149-57. doi: 10.1038/leu.2011.196. Epub 2011 Jul 29. PMID 21799510
- [Background] Kumar SK, Rajkumar V, Kyle RA, van Duin M, Sonneveld P, Mateos MV, Gay F, Anderson KC. Multiple myeloma. Nat Rev Dis Primers. 2017 Jul 20;3:17046. doi: 10.1038/nrdp.2017.46. PMID 28726797
- [Background] Kumar SK, Callander NS, Alsina M, Atanackovic D, Biermann JS, Castillo J, Chandler JC, Costello C, Faiman M, Fung HC, Godby K, Hofmeister C, Holmberg L, Holstein S, Huff CA, Kang Y, Kassim A, Liedtke M, Malek E, Martin T, Neppalli VT, Omel J, Raje N, Singhal S, Somlo G, Stockerl-Goldstein K, Weber D, Yahalom J, Kumar R, Shead DA. NCCN Guidelines Insights: Multiple Myeloma, Version 3.2018. J Natl Compr Canc Netw. 2018 Jan;16(1):11-20. doi: 10.6004/jnccn.2018.0002. PMID 29295877
- [Background] Kumar S, Paiva B, Anderson KC, Durie B, Landgren O, Moreau P, Munshi N, Lonial S, Blade J, Mateos MV, Dimopoulos M, Kastritis E, Boccadoro M, Orlowski R, Goldschmidt H, Spencer A, Hou J, Chng WJ, Usmani SZ, Zamagni E, Shimizu K, Jagannath S, Johnsen HE, Terpos E, Reiman A, Kyle RA, Sonneveld P, Richardson PG, McCarthy P, Ludwig H, Chen W, Cavo M, Harousseau JL, Lentzsch S, Hillengass J, Palumbo A, Orfao A, Rajkumar SV, Miguel JS, Avet-Loiseau H. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016 Aug;17(8):e328-e346. doi: 10.1016/S1470-2045(16)30206-6. PMID 27511158
- [Background] Kyprolis. [Package Insert]. Thousand Oaks, California, United States: Amgen. Available from: https://www.pi.amgen.com/~/media/amgen/repositorysites/pi-amgen- com/kyprolis/kyprolis_pi.pdf.
- [Background] Kyprolis. [Summary of Product Characteristics]. Breda, Netherlands: Amgen Europe BV. Available from: https://www.ema.europa.eu/en/documents/product-information/kyprolis-epar- product-information_en.pdf.
- [Background] Laabi Y, Gras MP, Brouet JC, Berger R, Larsen CJ, Tsapis A. The BCMA gene, preferentially expressed during B lymphoid maturation, is bidirectionally transcribed. Nucleic Acids Res. 1994 Apr 11;22(7):1147-54. doi: 10.1093/nar/22.7.1147. PMID 8165126
- [Background] Larocca A, Mina R, Gay F, Bringhen S, Boccadoro M. Emerging drugs and combinations to treat multiple myeloma. Oncotarget. 2017 Jul 15;8(36):60656-60672. doi: 10.18632/oncotarget.19269. eCollection 2017 Sep 1. PMID 28948001
- [Background] Landgren O, Devlin S, Boulad M, Mailankody S. Role of MRD status in relation to clinical outcomes in newly diagnosed multiple myeloma patients: a meta-analysis. Bone Marrow Transplant. 2016 Dec;51(12):1565-1568. doi: 10.1038/bmt.2016.222. Epub 2016 Sep 5. PMID 27595280
- [Background] Lokhorst HM, Plesner T, Laubach JP, Nahi H, Gimsing P, Hansson M, Minnema MC, Lassen U, Krejcik J, Palumbo A, van de Donk NW, Ahmadi T, Khan I, Uhlar CM, Wang J, Sasser AK, Losic N, Lisby S, Basse L, Brun N, Richardson PG. Targeting CD38 with Daratumumab Monotherapy in Multiple Myeloma. N Engl J Med. 2015 Sep 24;373(13):1207-19. doi: 10.1056/NEJMoa1506348. Epub 2015 Aug 26. PMID 26308596
- [Background] Lonial S, Dimopoulos M, Palumbo A, White D, Grosicki S, Spicka I, Walter-Croneck A, Moreau P, Mateos MV, Magen H, Belch A, Reece D, Beksac M, Spencer A, Oakervee H, Orlowski RZ, Taniwaki M, Rollig C, Einsele H, Wu KL, Singhal A, San-Miguel J, Matsumoto M, Katz J, Bleickardt E, Poulart V, Anderson KC, Richardson P; ELOQUENT-2 Investigators. Elotuzumab Therapy for Relapsed or Refractory Multiple Myeloma. N Engl J Med. 2015 Aug 13;373(7):621-31. doi: 10.1056/NEJMoa1505654. Epub 2015 Jun 2. PMID 26035255
- [Background] Lonial S, van de Donk N, Popat R, Zonder JA, Minnema MC, Larsen J, et al. First clinical (phase 1b/2a) study of iberdomide (CC-220; IBER), a CELMoD, in combination with dexamethasone (DEX) in patients (pts) with relapsed/refractory multiple myeloma (RRMM). J Clin Oncol. 2019;37(Suppl 15):8006.
- [Background] Lopez-Girona A, Mendy D, Ito T, Miller K, Gandhi AK, Kang J, Karasawa S, Carmel G, Jackson P, Abbasian M, Mahmoudi A, Cathers B, Rychak E, Gaidarova S, Chen R, Schafer PH, Handa H, Daniel TO, Evans JF, Chopra R. Cereblon is a direct protein target for immunomodulatory and antiproliferative activities of lenalidomide and pomalidomide. Leukemia. 2012 Nov;26(11):2326-35. doi: 10.1038/leu.2012.119. Epub 2012 May 3. PMID 22552008
- [Background] Lu G, Middleton RE, Sun H, Naniong M, Ott CJ, Mitsiades CS, Wong KK, Bradner JE, Kaelin WG Jr. The myeloma drug lenalidomide promotes the cereblon-dependent destruction of Ikaros proteins. Science. 2014 Jan 17;343(6168):305-9. doi: 10.1126/science.1244917. Epub 2013 Nov 29. PMID 24292623
- [Background] Ludwig H, Miguel JS, Dimopoulos MA, Palumbo A, Garcia Sanz R, Powles R, Lentzsch S, Ming Chen W, Hou J, Jurczyszyn A, Romeril K, Hajek R, Terpos E, Shimizu K, Joshua D, Hungria V, Rodriguez Morales A, Ben-Yehuda D, Sondergeld P, Zamagni E, Durie B. International Myeloma Working Group recommendations for global myeloma care. Leukemia. 2014 May;28(5):981-92. doi: 10.1038/leu.2013.293. Epub 2013 Oct 9. PMID 24177258
- [Background] Matyskiela ME, Zhang W, Man HW, Muller G, Khambatta G, Baculi F, Hickman M, LeBrun L, Pagarigan B, Carmel G, Lu CC, Lu G, Riley M, Satoh Y, Schafer P, Daniel TO, Carmichael J, Cathers BE, Chamberlain PP. A Cereblon Modulator (CC-220) with Improved Degradation of Ikaros and Aiolos. J Med Chem. 2018 Jan 25;61(2):535-542. doi: 10.1021/acs.jmedchem.6b01921. Epub 2017 Apr 20. PMID 28425720
- [Background] Mateos MV, Nahi H, Legiec W, Grosicki S, Vorobyev V, Spicka I, et al. Efficacy and safety of the randomized, open-label, non-inferiority, phase 3 study of subcutaneous (SC) versus intravenous (IV) daratumumab (DARA) administration in patients (pts) with relapsed or refractory multiple myeloma (RRMM): COLUMBA. J Clin Oncol. 2019; 37(Suppl 15):8005.
- [Background] Maus MV, Grupp SA, Porter DL, June CH. Antibody-modified T cells: CARs take the front seat for hematologic malignancies. Blood. 2014 Apr 24;123(17):2625-35. doi: 10.1182/blood-2013-11-492231. Epub 2014 Feb 27. PMID 24578504
- [Background] Moreau P, Masszi T, Grzasko N, Bahlis NJ, Hansson M, Pour L, Sandhu I, Ganly P, Baker BW, Jackson SR, Stoppa AM, Simpson DR, Gimsing P, Palumbo A, Garderet L, Cavo M, Kumar S, Touzeau C, Buadi FK, Laubach JP, Berg DT, Lin J, Di Bacco A, Hui AM, van de Velde H, Richardson PG; TOURMALINE-MM1 Study Group. Oral Ixazomib, Lenalidomide, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2016 Apr 28;374(17):1621-34. doi: 10.1056/NEJMoa1516282. PMID 27119237
- [Background] Moreau P, San Miguel J, Sonneveld P, Mateos MV, Zamagni E, Avet-Loiseau H, Hajek R, Dimopoulos MA, Ludwig H, Einsele H, Zweegman S, Facon T, Cavo M, Terpos E, Goldschmidt H, Attal M, Buske C; ESMO Guidelines Committee. Multiple myeloma: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv52-iv61. doi: 10.1093/annonc/mdx096. No abstract available. PMID 28453614
- [Background] Moreau P, Mateos MV, Berenson JR, Weisel K, Lazzaro A, Song K, Dimopoulos MA, Huang M, Zahlten-Kumeli A, Stewart AK. Once weekly versus twice weekly carfilzomib dosing in patients with relapsed and refractory multiple myeloma (A.R.R.O.W.): interim analysis results of a randomised, phase 3 study. Lancet Oncol. 2018 Jul;19(7):953-964. doi: 10.1016/S1470-2045(18)30354-1. Epub 2018 Jun 1. PMID 29866475
- [Background] Munshi NC, Longo DL, Anderson KC. Plasma cell disorders In: Oncology and Hematology 2012; Chapter 111: p. 936-944.
- [Background] Noone AM, Howlader N, Krapcho M, Miller D, Brest A, Yu M, Ruhl J, Tatalovich Z, Mariotto A, Lewis DR, Chen HS, Feuer EJ, Cronin KA (eds). SEER Cancer Statistics Review, 1975-2015, National Cancer Institute. Bethesda, MD, https://seer.cancer.gov/csr/1975_2015/, based on November 2017 SEER data submission, posted to the SEER web site, April 2018.
- [Background] Novak AJ, Darce JR, Arendt BK, Harder B, Henderson K, Kindsvogel W, Gross JA, Greipp PR, Jelinek DF. Expression of BCMA, TACI, and BAFF-R in multiple myeloma: a mechanism for growth and survival. Blood. 2004 Jan 15;103(2):689-94. doi: 10.1182/blood-2003-06-2043. Epub 2003 Sep 25. PMID 14512299
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Paiva B, van Dongen JJ, Orfao A. New criteria for response assessment: role of minimal residual disease in multiple myeloma. Blood. 2015 May 14;125(20):3059-68. doi: 10.1182/blood-2014-11-568907. Epub 2015 Apr 2. PMID 25838346
- [Background] Palumbo A, Anderson K. Multiple myeloma. N Engl J Med. 2011 Mar 17;364(11):1046-60. doi: 10.1056/NEJMra1011442. No abstract available. PMID 21410373
- [Background] Palumbo A, Bringhen S, Mateos MV, Larocca A, Facon T, Kumar SK, Offidani M, McCarthy P, Evangelista A, Lonial S, Zweegman S, Musto P, Terpos E, Belch A, Hajek R, Ludwig H, Stewart AK, Moreau P, Anderson K, Einsele H, Durie BG, Dimopoulos MA, Landgren O, San Miguel JF, Richardson P, Sonneveld P, Rajkumar SV. Geriatric assessment predicts survival and toxicities in elderly myeloma patients: an International Myeloma Working Group report. Blood. 2015 Mar 26;125(13):2068-74. doi: 10.1182/blood-2014-12-615187. Epub 2015 Jan 27. PMID 25628469
- [Background] Palumbo A, Chanan-Khan A, Weisel K, Nooka AK, Masszi T, Beksac M, Spicka I, Hungria V, Munder M, Mateos MV, Mark TM, Qi M, Schecter J, Amin H, Qin X, Deraedt W, Ahmadi T, Spencer A, Sonneveld P; CASTOR Investigators. Daratumumab, Bortezomib, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2016 Aug 25;375(8):754-66. doi: 10.1056/NEJMoa1606038. PMID 27557302
- [Background] Raje N, Hege K, Kochenderfer JN. Anti-BCMA CAR T-Cell Therapy in Multiple Myeloma. Reply. N Engl J Med. 2019 Jul 18;381(3):e6. doi: 10.1056/NEJMc1907520. No abstract available. PMID 31314982
- [Background] Palumbo A, Rajkumar SV, San Miguel JF, Larocca A, Niesvizky R, Morgan G, Landgren O, Hajek R, Einsele H, Anderson KC, Dimopoulos MA, Richardson PG, Cavo M, Spencer A, Stewart AK, Shimizu K, Lonial S, Sonneveld P, Durie BG, Moreau P, Orlowski RZ. International Myeloma Working Group consensus statement for the management, treatment, and supportive care of patients with myeloma not eligible for standard autologous stem-cell transplantation. J Clin Oncol. 2014 Feb 20;32(6):587-600. doi: 10.1200/JCO.2013.48.7934. Epub 2014 Jan 13. PMID 24419113
- [Background] Plesner T, Arkenau HT, Gimsing P, Krejcik J, Lemech C, Minnema MC, Lassen U, Laubach JP, Palumbo A, Lisby S, Basse L, Wang J, Sasser AK, Guckert ME, de Boer C, Khokhar NZ, Yeh H, Clemens PL, Ahmadi T, Lokhorst HM, Richardson PG. Phase 1/2 study of daratumumab, lenalidomide, and dexamethasone for relapsed multiple myeloma. Blood. 2016 Oct 6;128(14):1821-1828. doi: 10.1182/blood-2016-07-726729. Epub 2016 Aug 16. PMID 27531679
- [Background] Pomalyst. [Package Insert]. Summit, NJ: Celgene Corporation. Available from: http://www.pomalyst.com/wp-content/uploads/2013/08/prescribing_information.pdf.
- [Background] Pulte D, Gondos A, Brenner H. Improvement in survival of older adults with multiple myeloma: results of an updated period analysis of SEER data. Oncologist. 2011;16(11):1600-3. doi: 10.1634/theoncologist.2011-0229. Epub 2011 Oct 3. PMID 21968047
- [Background] Rajkumar SV. Multiple myeloma: 2011 update on diagnosis, risk-stratification, and management. Am J Hematol. 2011 Jan;86(1):57-65. doi: 10.1002/ajh.21913. PMID 21181954
- [Background] Rajkumar SV, Kumar S. Multiple Myeloma: Diagnosis and Treatment. Mayo Clin Proc. 2016 Jan;91(1):101-19. doi: 10.1016/j.mayocp.2015.11.007. PMID 26763514
- [Background] Revlimid. [Package Insert]. Summit, NJ: Celgene Corporation. Available from: http://www.revlimid.com/.
- [Background] Revlimid ™. [Summary of Product Characteristics]. Uxbridge, United Kingdom: Celgene Europe Ltd. Available from: http://www.ema.europa.eu/docs/en_GB/document_library/EPAR_- _Product_Information/human/000717/WC500056018.pdf.
- [Background] Richardson PG, Siegel DS, Vij R, Hofmeister CC, Baz R, Jagannath S, Chen C, Lonial S, Jakubowiak A, Bahlis N, Song K, Belch A, Raje N, Shustik C, Lentzsch S, Lacy M, Mikhael J, Matous J, Vesole D, Chen M, Zaki MH, Jacques C, Yu Z, Anderson KC. Pomalidomide alone or in combination with low-dose dexamethasone in relapsed and refractory multiple myeloma: a randomized phase 2 study. Blood. 2014 Mar 20;123(12):1826-32. doi: 10.1182/blood-2013-11-538835. Epub 2014 Jan 13. PMID 24421329
- [Background] Richardson P, Oriol Rocafiguera A, Beksac M, Marina Liberati A, Galli M, Schjesvold F, et al. Pomalidomide (POM), bortezomib, and low-dose dexamethasone (PVd) vs bortezomib and low-dose dexamethasone (Vd) in lenalidomide (LEN)-exposed patients (pts) with relapsed or refractory multiple myeloma (RRMM): Phase 3 OPTIMISMM trial. J Clin Oncol. 2018 May 20;36(Suppl):8001.
- [Background] Richardson PG, Barlogie B, Berenson J, Singhal S, Jagannath S, Irwin D, Rajkumar SV, Srkalovic G, Alsina M, Alexanian R, Siegel D, Orlowski RZ, Kuter D, Limentani SA, Lee S, Hideshima T, Esseltine DL, Kauffman M, Adams J, Schenkein DP, Anderson KC. A phase 2 study of bortezomib in relapsed, refractory myeloma. N Engl J Med. 2003 Jun 26;348(26):2609-17. doi: 10.1056/NEJMoa030288. PMID 12826635
- [Background] Richardson PG, Barlogie B, Berenson J, Singhal S, Jagannath S, Irwin DH, Rajkumar SV, Srkalovic G, Alsina M, Anderson KC. Extended follow-up of a phase II trial in relapsed, refractory multiple myeloma:: final time-to-event results from the SUMMIT trial. Cancer. 2006 Mar 15;106(6):1316-9. doi: 10.1002/cncr.21740. PMID 16470606
- [Background] Richardson PG, Jagannath S, Jakubowiak AJ, Lonial S, Raje N, Alsina M, et al. Phase II trial of lenalidomide bortezomib and dexamethasone in patients (pts) with relapsed and relapsed/refractory multiple myeloma (MM): Updated efficacy and safety data after >2 years of follow-up. Blood. 2010;116(Suppl 1):3049.
- [Background] Richardson PG, Blood E, Mitsiades CS, Jagannath S, Zeldenrust SR, Alsina M, Schlossman RL, Rajkumar SV, Desikan KR, Hideshima T, Munshi NC, Kelly-Colson K, Doss D, McKenney ML, Gorelik S, Warren D, Freeman A, Rich R, Wu A, Olesnyckyj M, Wride K, Dalton WS, Zeldis J, Knight R, Weller E, Anderson KC. A randomized phase 2 study of lenalidomide therapy for patients with relapsed or relapsed and refractory multiple myeloma. Blood. 2006 Nov 15;108(10):3458-64. doi: 10.1182/blood-2006-04-015909. Epub 2006 Jul 13. PMID 16840727
- [Background] Richardson PG, Siegel DS, Vij R, Hofmeister CC, Jagannath S, Chen C, et al. Randomized open label phase 1/2 study of pomalidomide (POM) alone or in combination with low-dose dexamethasone (LoDex) in patients (Pts) with relapsed and refractory multiple myeloma who have received prior treatment that includes lenalidomide (LEN) and bortezomib (BORT): Phase 2 results. Blood. 2011;118(Suppl 1):634.
- [Background] Richardson PG, Sonneveld P, Schuster M, Irwin D, Stadtmauer E, Facon T, Harousseau JL, Ben-Yehuda D, Lonial S, Goldschmidt H, Reece D, Miguel JS, Blade J, Boccadoro M, Cavenagh J, Alsina M, Rajkumar SV, Lacy M, Jakubowiak A, Dalton W, Boral A, Esseltine DL, Schenkein D, Anderson KC. Extended follow-up of a phase 3 trial in relapsed multiple myeloma: final time-to-event results of the APEX trial. Blood. 2007 Nov 15;110(10):3557-60. doi: 10.1182/blood-2006-08-036947. Epub 2007 Aug 9. PMID 17690257
- [Background] Richardson PG, Sonneveld P, Schuster MW, Irwin D, Stadtmauer EA, Facon T, Harousseau JL, Ben-Yehuda D, Lonial S, Goldschmidt H, Reece D, San-Miguel JF, Blade J, Boccadoro M, Cavenagh J, Dalton WS, Boral AL, Esseltine DL, Porter JB, Schenkein D, Anderson KC; Assessment of Proteasome Inhibition for Extending Remissions (APEX) Investigators. Bortezomib or high-dose dexamethasone for relapsed multiple myeloma. N Engl J Med. 2005 Jun 16;352(24):2487-98. doi: 10.1056/NEJMoa043445. PMID 15958804
- [Background] Sadelain M, Brentjens R, Riviere I. The basic principles of chimeric antigen receptor design. Cancer Discov. 2013 Apr;3(4):388-98. doi: 10.1158/2159-8290.CD-12-0548. Epub 2013 Apr 2. PMID 23550147
- [Background] San-Miguel JF, Hungria VT, Yoon SS, Beksac M, Dimopoulos MA, Elghandour A, Jedrzejczak WW, Gunther A, Nakorn TN, Siritanaratkul N, Corradini P, Chuncharunee S, Lee JJ, Schlossman RL, Shelekhova T, Yong K, Tan D, Numbenjapon T, Cavenagh JD, Hou J, LeBlanc R, Nahi H, Qiu L, Salwender H, Pulini S, Moreau P, Warzocha K, White D, Blade J, Chen W, de la Rubia J, Gimsing P, Lonial S, Kaufman JL, Ocio EM, Veskovski L, Sohn SK, Wang MC, Lee JH, Einsele H, Sopala M, Corrado C, Bengoudifa BR, Binlich F, Richardson PG. Panobinostat plus bortezomib and dexamethasone versus placebo plus bortezomib and dexamethasone in patients with relapsed or relapsed and refractory multiple myeloma: a multicentre, randomised, double-blind phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1195-206. doi: 10.1016/S1470-2045(14)70440-1. Epub 2014 Sep 18. PMID 25242045
- [Background] Miguel JS, Weisel K, Moreau P, Lacy M, Song K, Delforge M, Karlin L, Goldschmidt H, Banos A, Oriol A, Alegre A, Chen C, Cavo M, Garderet L, Ivanova V, Martinez-Lopez J, Belch A, Palumbo A, Schey S, Sonneveld P, Yu X, Sternas L, Jacques C, Zaki M, Dimopoulos M. Pomalidomide plus low-dose dexamethasone versus high-dose dexamethasone alone for patients with relapsed and refractory multiple myeloma (MM-003): a randomised, open-label, phase 3 trial. Lancet Oncol. 2013 Oct;14(11):1055-1066. doi: 10.1016/S1470-2045(13)70380-2. Epub 2013 Sep 3. PMID 24007748
- [Background] Sehgal K, Das R, Zhang L, Verma R, Deng Y, Kocoglu M, Vasquez J, Koduru S, Ren Y, Wang M, Couto S, Breider M, Hansel D, Seropian S, Cooper D, Thakurta A, Yao X, Dhodapkar KM, Dhodapkar MV. Clinical and pharmacodynamic analysis of pomalidomide dosing strategies in myeloma: impact of immune activation and cereblon targets. Blood. 2015 Jun 25;125(26):4042-51. doi: 10.1182/blood-2014-11-611426. Epub 2015 Apr 13. PMID 25869284
- [Background] Siegel DS, Dimopoulos MA, Ludwig H, Facon T, Goldschmidt H, Jakubowiak A, San-Miguel J, Obreja M, Blaedel J, Stewart AK. Improvement in Overall Survival With Carfilzomib, Lenalidomide, and Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma. J Clin Oncol. 2018 Mar 10;36(8):728-734. doi: 10.1200/JCO.2017.76.5032. Epub 2018 Jan 17. PMID 29341834
- [Background] Sonneveld P, Avet-Loiseau H, Lonial S, Usmani S, Siegel D, Anderson KC, Chng WJ, Moreau P, Attal M, Kyle RA, Caers J, Hillengass J, San Miguel J, van de Donk NW, Einsele H, Blade J, Durie BG, Goldschmidt H, Mateos MV, Palumbo A, Orlowski R. Treatment of multiple myeloma with high-risk cytogenetics: a consensus of the International Myeloma Working Group. Blood. 2016 Jun 16;127(24):2955-62. doi: 10.1182/blood-2016-01-631200. Epub 2016 Mar 21. PMID 27002115
- [Background] Stewart AK, Rajkumar SV, Dimopoulos MA, Masszi T, Spicka I, Oriol A, Hajek R, Rosinol L, Siegel DS, Mihaylov GG, Goranova-Marinova V, Rajnics P, Suvorov A, Niesvizky R, Jakubowiak AJ, San-Miguel JF, Ludwig H, Wang M, Maisnar V, Minarik J, Bensinger WI, Mateos MV, Ben-Yehuda D, Kukreti V, Zojwalla N, Tonda ME, Yang X, Xing B, Moreau P, Palumbo A; ASPIRE Investigators. Carfilzomib, lenalidomide, and dexamethasone for relapsed multiple myeloma. N Engl J Med. 2015 Jan 8;372(2):142-52. doi: 10.1056/NEJMoa1411321. Epub 2014 Dec 6. PMID 25482145
- [Background] Tai YT, Acharya C, An G, Moschetta M, Zhong MY, Feng X, Cea M, Cagnetta A, Wen K, van Eenennaam H, van Elsas A, Qiu L, Richardson P, Munshi N, Anderson KC. APRIL and BCMA promote human multiple myeloma growth and immunosuppression in the bone marrow microenvironment. Blood. 2016 Jun 23;127(25):3225-36. doi: 10.1182/blood-2016-01-691162. Epub 2016 Apr 28. PMID 27127303
- [Background] Thalidomide. [Summary of Product Characteristics]. Uxbridge, United Kingdom: Celgene Europe Ltd. Available from: https://www.ema.europa.eu/en/documents/product- information/thalidomide-celgene-epar-product-information_en.pdf.
- [Background] Thalomid. [Package Insert]. Summit, NJ: Celgene Corporation. Available from: http://www.celgene.com/content/uploads/thalomid-pi.pdf.
- [Background] Topp MS, Duell J, Zugmaier G, Attal M, Moreau P, Langer C, et al. Evaluation of AMG 420, an anti-BCMA bispecific T-cell engager (BiTE) immunotherapy, in R/R multiple myeloma (MM) patients: Updated results of a first-in-human (FIH) phase I dose escalation study. J Clin Oncol. 2019 May 26;37(Suppl 15):8007.
- [Background] van de Velde H, Londhe A, Ataman O, Johns HL, Hill S, Landers E, Berlin JA. Association between complete response and outcomes in transplant-eligible myeloma patients in the era of novel agents. Eur J Haematol. 2017 Mar;98(3):269-279. doi: 10.1111/ejh.12829. Epub 2016 Dec 17. PMID 27859769
- [Background] Velcade. [Package Insert]. Cambridge, MA: Millennium Pharmaceuticals. Available from: http://www.velcade.com/files/PDFs/VELCADE_PRESCRIBING_INFORMATION.pdf. Accessed on 02/16/2018.
- [Background] Velcade. [Summary of Product Characteristics]. Beerse, Belgium: Janssen-Cilag International NV. Available from: https://www.ema.europa.eu/en/documents/product-information/velcade- epar-product-information_en.pdf.
- [Background] Willenbacher E, Balog A, Willenbacher W. Short overview on the current standard of treatment in newly diagnosed multiple myeloma. Memo. 2018;11(1):59-64. doi: 10.1007/s12254-018-0383-3. Epub 2018 Feb 21. PMID 29606980
- [Background] Xu Y, Zhang M, Ramos CA, Durett A, Liu E, Dakhova O, Liu H, Creighton CJ, Gee AP, Heslop HE, Rooney CM, Savoldo B, Dotti G. Closely related T-memory stem cells correlate with in vivo expansion of CAR.CD19-T cells and are preserved by IL-7 and IL-15. Blood. 2014 Jun 12;123(24):3750-9. doi: 10.1182/blood-2014-01-552174. Epub 2014 Apr 29. PMID 24782509
- [Background] Yang Y, Shaffer AL 3rd, Emre NC, Ceribelli M, Zhang M, Wright G, Xiao W, Powell J, Platig J, Kohlhammer H, Young RM, Zhao H, Yang Y, Xu W, Buggy JJ, Balasubramanian S, Mathews LA, Shinn P, Guha R, Ferrer M, Thomas C, Waldmann TA, Staudt LM. Exploiting synthetic lethality for the therapy of ABC diffuse large B cell lymphoma. Cancer Cell. 2012 Jun 12;21(6):723-37. doi: 10.1016/j.ccr.2012.05.024. PMID 22698399
- [Background] Yong K, Delforge M, Driessen C, Fink L, Flinois A, Gonzalez-McQuire S, Safaei R, Karlin L, Mateos MV, Raab MS, Schoen P, Cavo M. Multiple myeloma: patient outcomes in real-world practice. Br J Haematol. 2016 Oct;175(2):252-264. doi: 10.1111/bjh.14213. Epub 2016 Jul 13. PMID 27411022
- [Background] Zhu YX, Braggio E, Shi CX, Bruins LA, Schmidt JE, Van Wier S, Chang XB, Bjorklund CC, Fonseca R, Bergsagel PL, Orlowski RZ, Stewart AK. Cereblon expression is required for the antimyeloma activity of lenalidomide and pomalidomide. Blood. 2011 Nov 3;118(18):4771-9. doi: 10.1182/blood-2011-05-356063. Epub 2011 Aug 22. PMID 21860026